CLINICAL TRIAL: NCT01190384
Title: Bean Consumption: A Pilot Study in Overweight Men and Women on Immuno-metabolic and Food Intake Endpoints
Brief Title: The Effect of Whole Beans on Inflammation and Satiety
Acronym: BEAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Illinois Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 201018072
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome; Inflammation; Antioxidants; Satiety; Fiber
MeSH Terms: conditions — Metabolic Syndrome; Inflammation | interventions — Dietary Fiber; Antioxidants; Grape Seed Extract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bean Soup (Experimental): Experimental soup with a high fiber content and ORAC value. The ORAC value is the Oxygen Radical Absorbance Capacity (ORAC) score which is a measure of the antioxidant levels of food and is expressed as Trolox Equivalents. The antioxidants in the soup are derived from beans.
  Interventions: Other: Bean Soup
- Couscous plus Fiber (Active Comparator): Soup with added fiber; has a low ORAC value. Subject serving is isocaloric to the experimental Bean soup.
  Interventions: Other: Couscous plus fiber
- Couscous plus Grape Seed Extract (Active Comparator): Control for ORAC value of the Bean soup; for examining the effect of fiber in the bean soup.
  Interventions: Dietary Supplement: Grape seed extract

INTERVENTIONS:
Other: Couscous plus fiber — Soup with added fiber to equal Bean soup. Subjects' serving size is isocaloric to the experimental Bean soup.
  Other Names: Non-active for antioxidants or fiber.
  Arms: Couscous plus Fiber
Dietary Supplement: Grape seed extract — 300 milligrams of grape seed extract in capsule form will be consumed with the low ORAC value soup.
  Other Names: Meganatural BP
  Arms: Couscous plus Grape Seed Extract
Other: Bean Soup — Experimental soup with a high fiber content and ORAC value. The ORAC value is the Oxygen Radical Absorbance Capacity (ORAC) score which is a measure of the antioxidant levels of food and is expressed as Trolox Equivalents. The antioxidants in the soup are derived from beans.
  Other Names: Whole black beans
  Arms: Bean Soup

SUMMARY:
Determine whether eating beans with a high fat meal will reduce the inflammatory response in people with the metabolic syndrome and increase feelings of satiety.

DETAILED DESCRIPTION:
Determine whether eating beans with a high fat meal will reduce the inflammatory response in people with the metabolic syndrome; thereby possibly postponing the diagnosis of diabetes or other chronic inflammatory diseases. These researchers are also interested in how consuming beans can affect the length of time a person stays full after a meal.

ELIGIBILITY:
Inclusion Criteria:

Men and Women 21 years old and older with metabolic syndrome

Exclusion Criteria:

1. Smokers
2. Female subjects who are pregnant or lactating
3. Subjects taking any medications that would interfere with outcomes of the study i.e. lipid lowering medications, anti-inflammatory drugs (i.e. ibuprofen), dietary supplements
4. Subjects with any known allergy or intolerance to foods involved in the study(cantaloupe, egg, dairy, wheat, beans, couscous, grape seed extract)
5. Subjects who are actively trying to lose weight
6. Subjects with unusual dietary habits (i.e. pica, anorexia nervosa, extreme food restriction, binging and/or purging disorders)
7. Subjects who are addicted to drugs or alcohol or who are <1 year recovery program
8. Subjects who present with significant psychiatric or neurological disturbances as determined by the primary investigator (i.e. uncontrolled bipolar disorder) These subjects will be referred to their primary care doctor for further care.
9. Subjects with documented atherosclerotic disease, inflammatory disease, diabetes mellitus (fasting blood sugar ≥126 mg/dl), uncontrolled hypertension (≥ 140/90mmHg), liver and kidney disease as identified by routine blood tests (chemistry panels). These subjects will be referred to their primary care doctor for further care.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-08; Primary Completion 2012-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Inflammation | 6 hours
  Measuring inflammatory markers after consumption of a high fat meal in conjunction with one of three soups. The three soups are: a bean soup high in fiber and antioxidants, a couscous soup high in fiber, and a couscous soup high in antioxidants.

SECONDARY OUTCOMES:
Satiety | 48 hours
  Measure subjects' perception of fullness during the 6 hour post-prandial testing period. Subjects will keep food records on the study day and day following to look for any longer effects on satiety as measured by food intake.

CONTACTS AND LOCATIONS:
Overall Officials: Chulani T Kappagoda, M.D., Ph.D., Principal Investigator — University of California, Davis
Locations (1):
- Ragle Human Nutrition Research Center, Davis, California, United States

REFERENCES:
- [Derived] Reverri EJ, Randolph JM, Kappagoda CT, Park E, Edirisinghe I, Burton-Freeman BM. Assessing beans as a source of intrinsic fiber on satiety in men and women with metabolic syndrome. Appetite. 2017 Nov 1;118:75-81. doi: 10.1016/j.appet.2017.07.013. Epub 2017 Jul 20. PMID 28735851